CLINICAL TRIAL: NCT04587843
Title: A Randomized Controlled Trial Evaluating the Effectiveness of Contrave (Naltrexone HCl and Bupropion HCl) in Patients Who Have Weight Recidivism Following Bariatric Surgery: Contrave Obesity Trials (COR) Weight Regain Study
Brief Title: A Trial Evaluating the Effectiveness of Contrave in Patients Who Have Weight Recidivism Following Bariatric Surgery
Acronym: COR-WR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Bausch Health, Canada Inc. (Unknown)
Responsible Party: Principal Investigator, Tony Chetty, Associate Professor Pathology and Molecular Medicine, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COR Weight Regain Study
Record Dates: First submitted 2020-10-05; First posted 2020-10-14 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Obesity
Keywords: weight recidivism; weight regain; inadequate weight loss
MeSH Terms: conditions — Obesity | interventions — bupropion hydrochloride, naltrexone hydrochoride drug combination

STUDY DESIGN:
Intervention Model Description: Parallel, randomized, double blind, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contrave 8mg/90mg Extended Release Tablet (Experimental): Group treated with Contrave Extended Release Tablets
  Interventions: Drug: Contrave 8Mg-90Mg Extended-Release Tablet
- Placebo (Placebo Comparator): Group given placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Contrave 8Mg-90Mg Extended-Release Tablet — Each Contrave Extended Release Tablet contains 8Mg of naltrexone HCl and 90Mg of bupropion HCl and will be administered orally. Total daily dose is 32Mg / 360Mg.
  Participants randomized to the treatment arm will be administered 4 Contrave tablets a day for 1 year (2 tablets taken twice a day).
  Other Names: naltrexone HCl/bupropion HCl
  Arms: Contrave 8mg/90mg Extended Release Tablet
Drug: Placebo — Placebo tablets will be administered orally. Participants randomized to the control arm will be administered 4 placebo tablets a day for 1 year (2 tablets, taken twice a day).
  Other Names: Inactive
  Arms: Placebo

SUMMARY:
Contrave (naltrexone HCl and bupropion HCl) extended-release tablet is an approved drug and indicated to be used with a low calorie diet and increased physical activity for chronic weight management in obese adults (BMI 30 Kg/m2 or greater) or overweight adults (BMI 27 Kg/m2 or greater) with at least one weight related condition such as hypertension or diabetes. It is unknown how many or which medical treatments for weight loss, such as Contrave work in the subjects who have had bariatric surgery.

The purpose of this study is to explore the effectiveness of Contrave combined with usual care (dietary and behaviour counselling) compared to placebo with usual care, in patients who have inadequate weight loss or significant weight regain following bariatric surgery.

DETAILED DESCRIPTION:
Obesity is associated with increased mortality and morbidity and represents a worldwide epidemic that is increasing in prevalence and remains a significant problem in Canada and a burden on our healthcare system. Maintaining long-term weight loss is the "Achilles' heel" of obesity therapy. Treatment for obesity with surgery is increasing because it has been shown to produce the best results for long-term weight loss and improving obesity related risk factors and diseases. But, these benefits are often reduced by inadequate weight loss or by weight regain in many patients after surgery.

Contrave (naltrexone HCl and bupropion HCl) extended-release tablet is an approved drug and indicated to be used with a low calorie diet and increased physical activity for chronic weight management in obese adults (BMI 30 Kg/m2 or greater) or overweight adults (BMI 27 Kg/m2 or greater) with at least one weight related condition such as hypertension or diabetes. It is unknown how many or which medical treatments for weight loss, such as Contrave work in the subjects who have had bariatric surgery.

This is a 1 year, phase 4, prospective, randomized, double-blind, placebo controlled study that will be conducted across multiple Bariatric Centres of Excellence (BCoE) in Ontario. Consenting participants will be randomly assigned to receive Contrave with usual care (dietary and behaviour counselling) or placebo with usual care. All subjects will also continue to receive usual care. The study includes several follow up visits to assess safety and treatment effects, some in person and others by telephone or video conferencing. Body weight, blood pressure, heart rate, waist circumference, lab tests, and subject completed questionnaires will be collected as part of usual care or for the study. Changes in medications and any possible side effects will also be monitored during the study.

To qualify, men and women must have had prior bariatric surgery (roux en-y gastric bypass or sleeve gastrectomy) at a surgical Center of Excellence within the Ontario Bariatric Network, and have inadequate weight loss or significant weight regain, based on the following OBN criteria:

1. < 10% total body weight (TBW) loss at 6 months or;
2. < 20% TBW loss at 12 months or;
3. Weight regain of > 25% of weight loss.

The aim of this study is to explore the effectiveness of Contrave combined with usual care (dietary and behaviour counselling) compared to placebo with usual care, in patients who have inadequate weight loss or significant weight regain following bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* >=18 years of age
* prior primary roux en-y gastric bypass (RYGB) or sleeve gastrectomy (SG) at a surgical Center of Excellence within the Ontario Bariatric Network (OBN)
* inadequate weight loss or significant weight regain based on the OBN criteria13, defined as one of the following:

  1. < 10% total body weight (TBW) loss at 6 months or;
  2. < 20% TBW loss at 12 months or;
  3. Weight regain of > 25% of weight loss.
* body Mass Index (BMI) of ≥ 30 Kg/m2 or ≥ 27 Kg/m2 and the presence of at least one weight related co-morbidity
* able and willing to provide signed informed consent

Exclusion Criteria:

* pregnancy, planned pregnancy in the next 18 months and or breastfeeding
* does not agree to use highly effective method of birth control if a woman of child bearing potential, for the duration of the study
* revisional bariatric procedure or duodenal switch
* simultaneous or planned use of other weight loss medication (e.g. Saxenda / Orlistat) or meal replacement products (e.g. Optifast)
* uncontrolled hypertension, severe hepatic impairment, end-stage renal disease, end stage cardiac disease
* myocardial infarction or stroke within 6 months prior to consent
* renal impairment defined as eGFR < 60
* seizure disorder or a history of seizures or following conditions that may predispose subjects to risk of seizure: history of head trauma, arteriovenous malformation, central nervous system tumor or infection, or a metabolic disorder that in opinion of the investigator may contraindicate treatment with Contrave and increase risk of seizure (e.g. hypoglycemia, hyponatremia)
* lifetime history of a suicide attempt or history of any suicidal behavior within the past month before entry into the trial
* history of major depressive disorder or a PHQ-9 (Patient Health Questionnaire-9) score of more than 15 within the last 2 years or history of other severe psychiatric disorders
* use of other bupropion-containing products (including, but not limited to, Wellbutrin, Wellbutrin SR, Wellbutrin XL, and Zyban), because the incidence of seizure is dose dependent
* current or prior diagnosis of bulimia or anorexia nervosa, because of a higher incidence of seizures
* chronic opioid or opiate agonist (eg, methadone) or partial agonists (eg, buprenorphine) use, or acute opiate withdrawal
* excessive use of alcohol or sedatives, addiction to cocaine or stimulants (street drugs), or withdrawal from sedatives
* patients undergoing an abrupt discontinuation of alcohol, benzodiazepines or other sedatives and antiepileptic drugs
* concomitant administration of monoamine oxidase inhibitors (MAOI). At least 14 days should elapse between discontinuation of a MAOI and initiation of treatment with Contrave
* concomitant administration of the antipsychotic thioridazine, since bupropion may inhibit thioridazine metabolism, thus causing an increase in thioridazine levels and a potential increased risk of thioridazine-related serious ventricular arrythmias and sudden death
* known hypersensitivity (or known allergic reaction) to the investigational product(s) or any of its ingredients including lactose
* current participation in another interventional clinical trial
* not able to complete subject reported, self administered questionnaires or cannot fully understand all instructions in English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in absolute weight (Kg) | Baseline to 12 months
  To determine the weight loss effect of Contrave with usual care compared to placebo with usual care, in a post-bariatric surgery population with weight loss failure.
Proportion of participants achieving 5 percent total weight loss | Baseline to 12 months
  To determine the weight loss effect of Contrave with usual care compared to placebo with usual care, in a post-bariatric surgery population with weight loss failure compared to a placebo with usual care.

SECONDARY OUTCOMES:
Change in Body Mass Index (BMI) (Kg/m2) | Baseline to 12 months
  To further determine effect of Contrave compared to placebo on BMI in a post-bariatric surgery population with weight loss failure.
Percentage total body weight loss (percentage TBWL) | Baseline to 12 months
  To determine effect of Contrave compared to placebo on weight loss in a post-bariatric surgery population with weight loss failure.
Proportion of participants losing at least 10 percent baseline weight at 12 months | Baseline to 12 months
  To further determine effect of Contrave compared to placebo on body weight in a post-bariatric surgery population with weight loss failure.
Percent change in HbA1c level | Baseline to 12 months
  To determine the effect of Contrave compared to placebo on HbA1c levels (laboratory blood test) as a measure of diabetic control in a post-bariatric surgery population with weight loss failure.
Change in blood pressure | Baseline to 12 months
  To determine the effect of Contrave compared to placebo on blood pressure and hypertension in a post-bariatric surgery population with weight loss failure.
Change in lipid profile | Baseline to 12 months
  To determine the effect of Contrave compared to placebo on lipid profile (total cholesterol, triglycerides, high density lipoprotein (HDL), low density lipoprotein (LDL)) in a post-bariatric surgery population with weight loss failure.
Changes in impulsivity behaviours from baseline as assessed by UPPS-P Impulsive Behaviour Scale (self administered questionnaire) | Baseline to 12 months
  To determine the effect of Contrave compared to placebo on impulsivity behaviours, in a post-bariatric surgery population with weight loss failure. Urgency, Premeditation (lack of), Perserverance (lack of), Sensation Seeking, Positive Urgency (UPPS-P Impulsive Behaviour Scale)
Changes in quality of life and health economic outcomes as measured with the EQ-5D-5L self administered questionnaire | Baseline to 12 months
  To determine the effect of Contrave compared to placebo on quality of life and health economic outcomes in a post-bariatric surgery population with weight loss failure.
Percentage of participants who are adherent to pharmacotherapy | Week 0 to Week 52
  To determine the tolerability of Contrave compared to placebo, in a post behaviour modification program setting.
Average number of days participants took investigational product (Contrave or placebo) | Week 0 to Week 52
  To determine the tolerability of Contrave compared to placebo, in a post behaviour modification program setting.
Change in diabetes medication requirements | Baseline to 12 months
  To determine the effect of Contrave compared to placebo on diabetic control in a post-bariatric surgery population with weight loss failure. If the patient is consuming diabetes medications, the diabetes medications will be documented during the study including any changes in medications, and any changes to dosing and frequency.
Change in hypertension (high blood pressure) medication requirements | Baseline to 12 months
  To determine the effect of Contrave compared to placebo on blood pressure and hypertension control in a post-bariatric surgery population with weight loss failure. If the patient is consuming medications for high blood pressure (hypertension), these medications will be documented during the study including any changes in medications, and any changes to dosing and frequency.
Change in lipid (cholesterol) medication requirements | Baseline to 12 months
  To determine the effect of Contrave compared to placebo on control of elevated total cholesterol, triglycerides and LDL with medication in a post-bariatric surgery population with weight loss failure. If the patient is consuming medications for elevated lipids (cholesterol, triglycerides LDL), these medications will be documented during the study including any changes in medications, and any changes to dosing and frequency.
Changes in eating behaviours from baseline as assessed by Eating Disorder Examination Questionnaire (EDE-Q 6.0) (self administered questionnaire) | Baseline to 12 months
  To determine the effect of Contrave compared to placebo on eating behaviours, in a post-bariatric surgery population with weight loss failure.
Changes in eating behaviours from baseline as assessed by Yale Food Addiction Scale (YFAS) (self administered questionnaire) | Baseline to 12 months
  To determine the effect of Contrave compared to placebo on eating behaviours, in a post-bariatric surgery population with weight loss failure.
Changes in food cravings from baseline as assessed by Favourite Food Craving Scale (FFCS) (self administered questionnaire) | Baseline to 12 months
  To determine the effect of Contrave compared to placebo on food cravings, in a post-bariatric surgery population with weight loss failure.
Changes in depression from baseline as assessed by Patient Health Questionnaire 9 (PHQ-9) (self administered questionnaire) | Baseline to 12 months
  To determine the effect of Contrave compared to placebo on depression and depressive problems, in a post-bariatric surgery population with weight loss failure.
Changes in risk of suicidality from baseline as assessed by the Columbia Suicide Severity Rating Scale (C-SSRS) | Baseline to 12 months
  To determine the effect of Contrave compared to placebo on risk of suicidality, in a post-bariatric surgery population with weight loss failure.

OTHER OUTCOMES:
Incidences of adverse events (AE) | Baseline to 12 months
  To determine the safety profile of Contrave in the setting of weight loss failure for post bariatric surgery patients.
Incidences of serious adverse events (SAE) | Baseline to 12 months
  To determine the safety profile of Contrave in the setting of weight loss failure for post bariatric surgery patients.
Number of participants discontinuing investigational product due to AE/SAEs | Baseline to 12 months
  To determine the tolerability profile of Contrave in the setting of weight loss failure for post bariatric surgery patients.

CONTACTS AND LOCATIONS:
Overall Officials: Aristithes G Doumouras, MD, Principal Investigator — St Joseph's Healthcare Hamilton / McMaster University
Locations (4):
- Canada (4):
  - Guelph General Hospital, Guelph, Ontario
  - St Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Humber River Hospital, North York, Ontario

IPD SHARING:
Plan to Share IPD: No